CLINICAL TRIAL: NCT03758248
Title: The Influence of Gene Polymorphism on Clinical Outcomes in Patients Undergoing PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Professor, Beijing Anzhen Hospital
Other Study IDs: Gene Polymorphism
Record Dates: First submitted 2018-11-15; First posted 2018-11-29 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Antiplatelet Therapy; CYP2C19 Polymorphism
Keywords: Genotype-guided therapy; CYP2C19 Polymorphism
MeSH Terms: interventions — Cytochrome P-450 CYP2C19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Gene polymorphism is measured by using whole blood in patients undergoing PCI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: CYP2C19 — The CYP2C19 enzyme plays a vital role in the two bioactivation steps of clopidogrel leading to lower (CYP2C19*17 carriers) or higher (CYP2C19*2 carriers) risk of major adverse cardiovascular events.

SUMMARY:
Dual antiplatelet therapy with aspirin and thienopyridines is an essential treatment in patients undergoing percutaneous coronary intervention (PCI). However, despite intensified antiplatelet treatment, some of the patients undergoing PCI develop thrombotic stent occlusion, suggesting incomplete platelet inhibition due to thienopyridine resistance. Some patients develop bleeding event because of the improper dosage and covariation. This observational study is designed for clarifying the Influence of gene polymorphism on clinical outcomes in patients undergoing PCI.

DETAILED DESCRIPTION:
Patients undergoing PCI who received dual antiplatelet therapy with both aspirin (100mg) and P2Y12 inhibitors in standard dosage were enrolled. Investigators examined plasma biomarkers for platelet activation and DNA in those patients, and then analyzed the CYP2C19 genetic polymorphism to examine the influence of this genetic variation on the several biomarkers for platelet activation and bleeding event.

ELIGIBILITY:
Inclusion Criteria:

1. The patients undergoing PCI
2. More than 18 years old
3. Treated with aspirin and P2Y12 inhibitors (clopidogrel or ticagrelor)

Exclusion Criteria:

Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PCI patients in Beijing Anzhen Hospital from August 2018 to August 2019
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Patients with treatment-related major bleeding event as assessed by the Bleeding Academic Research Consortium (BARC) bleeding criteria | up to 24 months
  The major bleeding event was a composite endpoint of BARC bleeding type 3 and 5), defined according to the BARC bleeding criteria, which was used widely in this field. BARC bleeding was defined as follows: BARC type 1, any bleeding that is not actionable; type 2, any overt, actionable sign of bleeding; type 3a, overt bleeding with a haemoglobin drop of 3-5 g/dL or any transfusion; type 3b, overt bleeding with a haemoglobin drop >5 g/dL, requiring vasopressors, surgical intervention, or due to cardiac tamponade; type 3c, any intracranial or intraocular bleeding; and finally type 5, any bleeding resulting in death (type 4 was coronary artery bypass graft-related bleeding, which was excluded). Investigator will get all the information through regular return visit and telephone follow-up after discharge.

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) | up to 24 months
  A composite of death, myocardial infarction, stroke, stent thrombosis, and ischemia-driven revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, PhD,MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided